CLINICAL TRIAL: NCT00418314
Title: FREEDOM - A Frequent Optimization Study Using the QuickOpt Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRD378
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Arrhythmias; Heart Failure
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QuickOpt (Treatment) (Experimental): Frequent optimization using QuickOpt to optimize the AV/PV and VV Delays.
  Interventions: Device: QuickOpt
- Control (Active Comparator): Empiric programming or one-time optimization using a non-IEGM method.
  Interventions: Device: Control

INTERVENTIONS:
Device: Control — Empiric programming or one-time optimization using a non-IEGM method.
  Arms: Control
Device: QuickOpt — Frequent optimization using QuickOpt to optimize AV/PV and VV delays.
  Arms: QuickOpt (Treatment)

SUMMARY:
The objective of this study is to demonstrate that frequent atrio-ventricular (AV/PV) and inter-ventricular (V-V) delay optimization using QuickOpt in patients with cardiac resynchronization therapy device results in improved clinical response over standard of care (i.e. empiric programming or one-time optimization using any non-intracardiac electrogram optimization methods).

DETAILED DESCRIPTION:
* This is a prospective, double-blinded, multicenter, randomized study
* Patient could be enrolled up to 2 weeks post CRT-D implant and are followed for 12 months post implant with follow-up visits at 3, 6, 9 and 12 months
* Patients will be randomized at enrollment to either Group 1 ("QuickOpt Group") or Group 2 ("Control Group").
* Group 1 - The patient's device is programmed to sequential biventricular pacing mode with AV/PV and VV delays optimized using QuickOpt. For Group 1 patients, optimization using QuickOpt is performed at enrollment, 3 month, 6 month, 9 month, 12 month and at any unscheduled follow-up visits.
* Group 2 - The patient's device is programmed to either simultaneous or sequential BiV pacing mode as per physician's discretion. The AV/PV and inter-ventricular (VV) delays could be programmed empirically or optimized using any non-IEGM based method as per sites standard of care. However, the Group 2 patients can be optimized only once within the first 4 weeks post implant. Any AV/PV and VV delay optimizations performed after 4 weeks post implant in Group 2 patients will be considered protocol deviations.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets current CRT-D indications and be implanted with a St. Jude Medical (SJM) CRT¬D device with VV timing and a compatible lead system.
* Patient has the ability to complete a 6-minute hall walk with the only limiting factor to be fatigue or shortness of breath.
* Patient has the ability to independently comprehend and complete a QOL questionnaire.

Exclusion Criteria:

* Patient has an epicardial ventricular lead system.
* Patient has the ability to walk ≥ 450 meters in 6 minutes
* Patient has limited intrinsic atrial activity (≤ 40 bpm).
* Patient has persistent or permanent atrial fibrillation (AF).
* Patient has a 2° or 3° heart block.
* Patient's life expectancy is less than 1 year.
* Patient is pregnant.
* Patient is on IV inotropic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1647 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Abraham, MD, Principal Investigator — Ohio State University, Columbus, OH, USA; Daniel Gras, MD, Principal Investigator — Nouvelles Cliniques Nantaises, Nantes, France
Locations (2):
- United States (2):
  - Cedars Sinai Hospital, Los Angeles, California
  - Ohio State Univeristy, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abraham WT, Gras D, Yu CM, Guzzo L, Gupta MS; FREEDOM Steering Committee. Rationale and design of a randomized clinical trial to assess the safety and efficacy of frequent optimization of cardiac resynchronization therapy: the Frequent Optimization Study Using the QuickOpt Method (FREEDOM) trial. Am Heart J. 2010 Jun;159(6):944-948.e1. doi: 10.1016/j.ahj.2010.02.034. PMID 20569704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QuickOpt (Treatment) | Control
Started | 817 | 830
Completed | 816 | 828
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Date of birth missing for 1 treatment patient and 1 control patient.
Groups:
- Total: Total of all reporting groups
Arm/Group | QuickOpt (Treatment) | Control | Total
Number analyzed (Participants) | 817 | 830 | 1647
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 307 | 340 | 647
  >=65 years | 510 | 490 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (11) | 66.7 (11) | 66.7 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 238 | 434
  Male | 621 | 592 | 1213
Region of Enrollment [Number; unit: participants]
  United States | 482 | 487 | 969
  Europe | 282 | 288 | 570
  Canada | 32 | 35 | 67
  Australia | 17 | 15 | 32
  Middle East | 3 | 4 | 7
  Southeast Asia | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Heart Failure Clinical Composite Score
Description: The clinical composite score classifies each randomized patient as improved, unchanged, or worse depending on the clinical response during and the clinical status at the end of the trial. Patients are considered improved if at the final visit they experienced a favorable change in NYHA functional class or in the patient global assessment (or both) but did not experience any major adverse clinical events during the course of the trial. Patients are considered worse if they experienced a major clinical event during the study duration or reported worsening of their NYHA class or global assessment at the final visit. Patients are considered unchanged if they are neither improved nor worse.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | QuickOpt (Treatment) | Control
Number analyzed (Participants) | 816 | 828
participants
  Improved | 551 | 559
  Unchanged | 76 | 86
  Worsened | 189 | 183

2. Secondary Outcome: All-cause, Cardiovascular and Heart Failure Mortality;
Time Frame: 12 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | QuickOpt (Treatment) | Control
Number analyzed (Participants) | 816 | 828
participants | 44 | 42

3. Secondary Outcome: All Cause, Cardiovascular and Heart Failure Hospitalization
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | QuickOpt (Treatment) | Control
Number analyzed (Participants) | 816 | 828
participants | 294 | 303

ADVERSE EVENTS:
Arm/Group | QuickOpt (Treatment) | Control
Serious Adverse Events (participants affected / at risk) | 120/816 | 111/828
Other Adverse Events (participants affected / at risk) | 184/816 | 177/828
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QuickOpt (Treatment) (N=816) | Control (N=828)
Coronary Angiogram (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmias (Cardiac disorders) | 11 (12) | 10 (10)
Cardiac Perforation (Cardiac disorders) | 2 (2) | 5 (5)
Thrombosis (Cardiac disorders) | 0 (0) | 3 (3)
Chest pain/MI (Cardiac disorders) | 7 (10) | 9 (10)
Coronary Sinus Dissection (Cardiac disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 8 (8) | 7 (7)
Device migration/malfunction (Cardiac disorders) | 0 (0) | 2 (3)
Elevated Pacing Thresholds (Cardiac disorders) | 10 (10) | 3 (3)
Erosion/Pocket Pain (Cardiac disorders) | 4 (4) | 2 (2)
Hematoma (Cardiac disorders) | 4 (4) | 7 (7)
Infection (Cardiac disorders) | 10 (10) | 14 (15)
Lead Dislodgment/Migration (Cardiac disorders) | 40 (45) | 35 (44)
Lead Fracture/Insulation Damage (Cardiac disorders) | 3 (3) | 0 (0)
Oversensing/Undersensing (Cardiac disorders) | 16 (18) | 8 (9)
Phrenic Nerve/Diaphragmatic Nerve Stimulation (Cardiac disorders) | 11 (12) | 6 (7)
Therapy for non-ventricular rhythm (Cardiac disorders) | 0 (0) | 3 (3)
Valve replacement (Cardiac disorders) | 0 (0) | 2 (2)
Other cardiac (Cardiac disorders) | 4 (4) | 3 (3)
Endocrine disorders (Endocrine disorders) | 2 (2) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
CVA/TIA (Nervous system disorders) | 2 (2) | 2 (2)
Neurologic other (Nervous system disorders) | 1 (1) | 1 (2)
DVT (Vascular disorders) | 3 (3) | 6 (9)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Respiratory other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QuickOpt (Treatment) (N=816) | Control (N=828)
Cardiopulmonary Arrest (Cardiac disorders) | 2 (2) | 4 (4)
Arrhythmias (Cardiac disorders) | 65 (83) | 55 (63)
Elevated Pacing Thresholds (Cardiac disorders) | 10 (13) | 3 (3)
Undersensing/Oversensing (Cardiac disorders) | 14 (16) | 11 (14)
Heart Failure (Cardiac disorders) | 61 (95) | 43 (63)
Hematoma (Cardiac disorders) | 7 (7) | 13 (13)
Infection (Cardiac disorders) | 4 (5) | 3 (3)
Lead Dislodgement/Migration (Cardiac disorders) | 14 (16) | 17 (20)
MI (Cardiac disorders) | 2 (2) | 5 (5)
Phrenic Nerve/Diaphragmatic Nerve Stimulation (Cardiac disorders) | 36 (47) | 30 (34)
Syncope (Nervous system disorders) | 8 (9) | 10 (10)
Therapy for non-ventricular rhythm (Cardiac disorders) | 5 (6) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications and presentations proposed by participating centers should be furnished to sponsor for review and comment 30 days (manuscripts) or 7 days (abstracts) prior to submission for publication. Sponsor reserves the right to deny submission of study results if based on data owned by sponsor.